CLINICAL TRIAL: NCT04126655
Title: A Randomised Phase II Study Investigating Two Doses of Arfolitixorin Compared to Calciumfolinate Together With 5- Fluorouracil on TS Inhibition in Tumour and Adjacent Hepatic Tissue for Patients With Liver Metastases From Colorectal Cancer
Brief Title: Modelle 001, TS-inhibition in Colorectal Liver Metastases Comparing Arfolitixorin and Calciumfolinate
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Isofol Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-005052-25
Record Dates: First submitted 2019-10-04; First posted 2019-10-15 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal cancer,; Liver metastases; 5-FU; Arfolitixorin; Calciumfolinate; TS-inhibtion
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: A total of 30 patients will be included in the study and will be equally randomised in three steps.
  In the first phase, six patients will receive a reduced dose 5-FU; 250 mg / m², of which three patients will be randomized to additional Calciumfolinate and three patients will be randomized to additional Arfolitixorin. P When all six patients have been followed up in the context of visits consultation, a clinical safety evaluation (SE) of all AE, and SAE will be performed by two independent physicians If the responsible physicians finds that it is safe that the study will continue, we intend to increase the dose of 5-FU 500 mg / m, after which additional 12 patients will be included.
  After inclusion of 6 patients receiving 5-FU 500 mg /m² in combination with Arfolitixorin in the dose of 30mg/m2 a dose adjustment will take place and the last 12 patients will be randomised to either Calciumfolinate 60 mg/m2 or Arfolitixorin 120 /m2.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomisation will be performed by a sealed envelope system. The randomisation envelopes are kept in a locked cabinet together with the randomisation list Two sets of code envelopes are prepared. The study personnel that will be responsible for study drug administration will have one set for the randomisation of patients and one set will be held by the investigator for emergency code breaking.
  The code envelopes are prepared for each patient and contain information about what treatment the patient should receive. The randomisation will be made by the study personnel responsible for the administration of the study drugs at the day of the surgery. The patients will be randomised in consecutive order. The date and time of randomisation should be recorded on the document followed by a signature of the person opening the envelope.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arfolitixorin. (Experimental): Drug: Arfolitixorin Drug: 5-FU Per operative i.v. bolus injection of Arfolitixorin in combination with 5-FU
  Interventions: Drug: Arfolitixorin
- Calciumfolinate. (Active Comparator): Drug: Calciumfolinate Drug: 5-FU Per operative i.v. bolus injection of Calciumfolinate in combination with 5-FU
  Interventions: Drug: Arfolitixorin

INTERVENTIONS:
Drug: Arfolitixorin — Per operative administration of 5-FU with Arfolitixorin or Calciumfolinate
  Other Names: Calciumfolinate

SUMMARY:
A study that is blinded to the patient and the investigator where the combination of Arfolitixorin + 5-FU is compared to Calciumfolinate + 5-FU. The patients will be randomised and will receive the above described combination as IV bolus injections, peroperatively in conjuction with collection of the first tissue sample.

A low dose (30 mg) and a high dose (120) mg of Arfolitixorin will be used in order to investigate the relation between dose of Arfolitixorin and TS-inhibition.

DETAILED DESCRIPTION:
Arfolitixorin ([6R] 5,10-methylenetetrahydrofolate) is a folate based biomodulator designed to replace leucovorin. Arfolitixorin is the key active metabolite of leucovorin (LV) and does in contrast to LV not require enzymatic metabolic activation. In clinical practice, LV is administered in the form of Calciumfolinate. A hypothesis is therefore that patients which are not capable of metabolizing LV could have a better antitumoral effect with Arfolitixorin administration. The antitumoural effect could be measured as inhibition of the enzyme thymidylate synthase, an enzyme essential for DNA synthesis.

Primary objective The primary objective is to compare the properties of Arfolitixorin and Calciumfolinate together with 5-fluorouracil (5-FU) on thymidylate synthase (TS) (i.e. measured as thymidylate synthase inhibition) in tumour and adjacent liver tissue in patients with liver metastases from colorectal cancer receiving a peroperative intravenous administration of Arfolitixorin or Calciumfolinate.

Secondary objectives To study safety in terms of adverse events and laboratory measurements; haematology and clinical chemistry.

To explore differences in pharmacokinetics of folates and folate metabolites in plasma.

To study gene expression in tumour and adjacent hepatic tissue and its correlation to tissue concentration.

To investigate the relation between the levels of deoxyuridine (dU) in plasma with the amount of TS inhibition in tumour tissue, in order to evaluate dU as a surrogate marker for TS-inhibition.

Study population:

Thirty adult patients with colorectal cancer and liver metastases, indicated for surgical removal will be randomised.

ELIGIBILITY:
Inclusion Criteria:

* 7.3.1 Inclusion criteria

  1. Patients must sign an informed consent document.
  2. At least two liver metastases secondary to CRC. Patients must have removable metastases amenable to surgery.
  3. Performance status of 0 to 2 on the Eastern Cooperative Oncology Group (ECOG). Performance Status scale. (See Protocol Attachment 1.)
  4. For women: Must be surgically sterile, postmenopausal, or compliant with a contraceptive regimen during and for 3 months after treatment. Fertile women must have a negative serum or urine pregnancy test (within 7 days before enrolment) and must not be lactating.
  5. For men: Must be surgically sterile or compliant with a contraceptive regimen during and for 3 months after treatment.
  6. Patient legally competent and able to communicate effectively with the study personnel as judged by the investigator.
  7. Patient likely to co-operate during the study.
  8. Patients must be at least 18 years of age.

     Exclusion Criteria:1.

     Concurrent administration of any other anti-tumour therapy minimum 3 weeks before surgery according to clinical practise.

  2. Treatment within the last 30 days with a drug/device that has not received regulatory approval for any indication at the time of study entry.

  3. Any intake of medication, which could influence folate, and vitamin B12 status, within 30 days of surgery.

  4. Serious concomitant systemic disorders (e.g., active infection including HIV, cardiac disease) that in the opinion of the investigator would compromise the patient's ability to complete the study.

  5. Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.

  6. Patients with a high risk of postoperative liver failure due to advanced liver metastatic load.

  7. Pregnancy. 8. History of significant neurological or mental disorder, including seizures or dementia.

  9. Presence of clinically relevant (i.e., detectable by physical examination) third-space fluid collection (e.g., ascites, pleural effusion) that cannot be controlled by drainage or other procedures prior to study entry.

  10. Known hypersensitivity to 5-FU and or Calciumfolinate/Arfolitixorin.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-05 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
TS inhibition i tumour tissue | Biopsies will be collected during liver surgery
  The primary objective is to compare the TS-inhibtion capacity of the combination Arfolitixorin/5-FU in contrast to Calciumfolinate/5-FU in tumour, adjacent liver parenchyma and plasma in patients with liver metastases from colorectal cancer
TS inhibition in adjacent liver parenchyma | Biopsies will be collected during live surgery
  The primary objective is to compare the TS-inhibtion capacity of the combination Arfolitixorin/5-FU in contrast to Calciumfolinate/5-FU in adjacent liver in patients with liver metastases from colorectal cancer
TS inhibition in plasma | Blood samples will be collected according to a sampling schedule during 24 hours after the bolus injection.
  The primary objective is to compare the TS-inhibtion capacity of the combination Arfolitixorin/5-FU in contrast to Calciumfolinate/5-FU in plasma in patients with liver metastases from colorectal cancer

CONTACTS AND LOCATIONS:
Overall Officials: Helena Taflin, MD, PhD, Principal Investigator — Vastra Gotaland Region
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No